CLINICAL TRIAL: NCT04999072
Title: Carbohydrate Antigen 19-9 Plus Carcinoembryonic Antigen for Prognosis in Colorectal Cancer
Brief Title: Carbohydrate Antigen 19-9 in Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Min Jung Kim, Assistant Professor, Seoul National University Hospital
Other Study IDs: SNUH_CA19-9
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Colectomy for colon cancer — Segmental or total colectomy was performed for colorectal cancer.

SUMMARY:
4,972 patients who underwent surgery for primary CRC between January 2004 and December 2015 at Seoul National University Hospital were retrospectively reviewed.

CA19-9 is a valuable prognostic and diagnostic marker for CRC when used adjunctively with CEA and can be a supplementary marker with CEA to improve sensitivity, especially with elevated preoperative CA19-9.

DETAILED DESCRIPTION:
Introduction: Carcinoembryonic antigen (CEA) is a main prognostic marker and can detect colorectal cancer (CRC) recurrence, but it has low sensitivity. Carbohydrate antigen 19-9 (CA19-9) can be used as a supplemental tumour marker along with CEA. This study investigated the utility of preoperative and follow-up serum CA19-9 assessment for CRC.

Materials and Methods: We retrospectively assessed 4,972 patients who underwent surgery for primary CRC between January 2004 and December 2015 at Seoul National University Hospital. Data on demographics, preoperative and follow-up CEA and CA19-9 levels, recurrence, and survival were obtained and analysed with respect to tumour marker levels to ascertain their prognostic and diagnostic values.

Results: The 5-year relapse-free survival rates were 72.2±0.8%, 52.5±2.2%, 55.5±3.2%, and 32.1±2.3% in the normal CEA and CA19-9, high CEA, high CA19-9, and high CEA and high CA19-9 groups, respectively (all p<0.001). Patients whose elevated CEA or CA19-9 reduced to normal had better survival outcomes than those with postoperatively elevated levels. Elevated follow-up CA19-9 and CEA levels were related to higher incidences of distant metastasis (CA19-9: 14.0% vs. 23.1%, p=0.004, CEA: 12.6% vs. 30.1%, p<0.001) but not with local recurrence. Combined follow-up CEA and CA19-9 increased the sensitivity for recurrence to 31.4%, with a 5% difference compared with CEA alone. In the subgroup with high preoperative CA19-9 levels, sensitivity increased by 18.2% overall.

Conclusion: CA19-9 is a valuable prognostic and diagnostic marker for CRC when used adjunctively with CEA and can be a supplementary marker with CEA to improve sensitivity, especially with elevated preoperative CA19-9.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgery for primary CRC between January 2004 and December 2015 at Seoul National University Hospital

Exclusion Criteria:

* The patients with missing data for preoperative and follow-up tumour markers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This single-centre retrospective study was based on the analysis of information from a prospectively maintained database of CRC in Seoul National University Hospital (SNUH CRC DB). Data were extracted from the SNUH CRC DB for patients who underwent surgery for primary CRC between January 2004 and December 2015 at our institution. The patients with missing data for preoperative and follow-up tumour markers were excluded from the analysis. This study was approved by the Institutional Review Board of Seoul National University Hospital (SNUH IRB; IRB no. 2007-014-1138). The approving authority waived the requirement for written informed consent owing to the retrospective study design.
Sampling Method: Non-Probability Sample
Enrollment: 4972 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Relapse free survival | 5-year
  Recurrence and death was the event for relapse free survival

CONTACTS AND LOCATIONS:
Overall Officials: Min Jung Kim, M.D., Principal Investigator — Seoul National University Hospital, Republic of Korea
Locations (1):
- Seoul National University Hospital, Seoul, Jongnogu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided